CLINICAL TRIAL: NCT03319121
Title: The Evaluation of Effectiveness Between Empirical and Guided Therapy for Unexplained Non-Cardiac Chest Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Yeong Yeh Lee, Professor Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14070265
Record Dates: First submitted 2017-10-18; First posted 2017-10-24 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Non Cardiac Chest Pain
Keywords: Non cardiac chest pain; Empirical therapy; Guided therapy
MeSH Terms: interventions — Dexlansoprazole

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated into either the empirical group or guided group for 8 weeks.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empirical therapy group (Experimental): Participants will be given extended release lansoprazole (Dexlansoprazole, Takeda Pharmaceuticals, Japan) 60 mg daily for 2 weeks
  Interventions: Drug: Empirical therapy group
- Guided therapy group (Experimental): Participants will be give Dexlansoprazole 30 mg daily for GERD, 60 mg daily for GERD with erosive esophagitis for 8 weeks and Theophylline SR 250 mg daily for functional chest pain for 4 weeks.
  Interventions: Drug: Guided therapy group

INTERVENTIONS:
Drug: Empirical therapy group — Receive extended release lansoprazole (Dexlansoprazole, Takeda Pharmaceuticals, Japan) 60 mg daily for 2 weeks.
  Other Names: Dexlansoprazole
  Arms: Empirical therapy group
Drug: Guided therapy group — Receive Dexlansoprazole 30 mg daily for GERD, 60 mg daily for GERD with erosive esophagitis for 8 weeks and Theophylline SR 250 mg daily for functional chest pain for 4 weeks.
  Other Names: Dexlansoprazole and/or Theophylline SR
  Arms: Guided therapy group

SUMMARY:
This is a prospective randomised clinical trial performed in a single center at Hospital Universiti Sains Malaysia (USM), Kelantan, Malaysia. Participants will be randomly allocated into either the empirical group or guided group for 8 weeks.The effectiveness in relieving chest pain (frequency and severity) will assessed after 2 weeks and 8 weeks of therapy with Gastroesophageal Reflux Disease Questionnaire (GERDQ) and Quality of Life Reflux and Dyspepsia (QOLRAD) questionnaire, and visual analogue scale (VAS) (score 1-10).

DETAILED DESCRIPTION:
Non-cardiac chest pain (NCCP) is very common in the general population but symptom alone or patient's characteristics do not adequately differentiate cardiac and esophageal cause. Cardiologists are usually consulted first to exclude life-threatening acute coronary syndrome. Tests that are performed to exclude ischemic heart disease include exercise stress test and the more invasive coronary angiography. A negative stress test or angiogram or the presence of mild blockage of a single vessel disease will usually be adequate to exclude significant ischemia as a cause for chest pain.

The next most important cause of unexplained chest pain would be gastro-esophageal reflux disease (GERD). GERD and its complications of Barrett's oesophagus and oesophageal adenocarcinoma have increased markedly in recent decades, not just in the developed countries but also in Asia. Although relatively less common among populations in Malaysia, there are data to suggest an increasing prevalence of reflux disease largely a result of obesity and increased intra-abdominal pressure.

Dexlansoprazole (Takeda Pharmaceuticals, Japan) is a novel dual delayed release system recently approved by the FDA for treatment of heartburn associated with non-erosive and erosive reflux disease. It is unknown if dexlansoprazole is effective as an empirical therapy for NCCP.

Another approach would be therapy guided by investigations including high resolution (HR) esophageal impedance manometry and 24-hour pH-impedance studies. Study of esophageal function has greatly evolved with the recent availability of high resolution multi-channel solid state manometer and impedance. Water swallows are commonly used in esophageal manometric studies to evaluate for peristaltic abnormalities. Esophageal pH monitoring does not detect all gastroesophageal reflux (GER) events but with the combination of impedance, this technique allows detection of GER of gas and acid or non-acid liquids. These tests would enable diagnosis of GERD and functional chest pain and thereby allow targeted therapy.

For treatment of GERD, dexlansoprazole is effective and for functional chest pain, nonspecific adenosine antagonist, theophylline is proven to improve symptoms in patient with hypersensitive esophagus. A selective serotonin reuptake inhibitor (SSRI) is also effective for functional chest pain , however it is not known if theophylline is more effective than any other SSRIs.It is unknown about the response rates based on the guided therapy approach compared to the empirical PPI therapy.

Therefore, the aim of the intervention is to evaluate the effectiveness of empirical therapy vs. guided therapy on symptoms unexplained non-cardiac chest pain.

ELIGIBILITY:
Inclusion Criteria: Participants with chest pain but normal angiogram or a negative stress test or normal electrocardiogram and cardiac enzyme.

Exclusion Criteria:

1. Participants with any medications that might affect the upper GI tract, previous surgeries of the upper GI tract and a negative endoscopic examination for peptic ulcer disease and upper GI tract malignancies
2. Participants with chronic, debilitating or life-threatening medical conditions and presence of overt psychiatric or psychological disturbances.

Ages: 18 Months to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Non-cardiac chest pain symptoms assessed by visual analog scale (VAS) | 8 weeks
  Visual analog scale (VAS) was used to assess the non-cardiac chest pain symptoms. VAS is a psychometric response scale. The scale has scores from 0 to 10 with 1 cm interval between scores and with 0 denotes no pain, 5 denote moderate pain and 10 denote the worst possible pain.

SECONDARY OUTCOMES:
Non-cardiac chest pain symptoms assessed by gastroesophageal reflux disease questionnaire (GERDQ) | 8 weeks
  Gastroesophageal reflux disease questionnaire (GERDQ) was used to assess the non-cardiac chest pain symptoms. GERDQ is a 6-item questionnaire developed for the diagnosis of GERD in a primary care setting. The total score of 0-8 is interpreted as less likely GERD and total score 9-18 is highly suggestive of GERD.
Non-cardiac chest pain symptoms assessed by quality of life in reflux and dyspepsia questionnaire (QOLRAD) | 8 weeks
  Quality of life in reflux and dyspepsia questionnaire (QOLRAD) was used to assess the non-cardiac chest pain symptoms. QOLRAD is a disease-specific questionnaire including 25 items combined into 5 dimensions: emotional distress, sleep disturbances, vitality, food/drinks problem and physical/social functioning. A seven-point graded Likert scale is used to rate the QOLRAD. Lower scores indicate a more severe impact on daily life and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Yeong Yeh Lee, MD, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospitial Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

REFERENCES:
- [Derived] Abdul Kadir NP, Ma ZF, Abdul Hafidz MI, Annamalai C, Jayaraman T, Hamid N, Norhasliza S, Abd Aziz A, Yusof Z, Lee H, Lee YY. Comparing Efficacy and Safety of Empirical vs. Guided Therapy for Non-cardiac Chest Pain: A Pragmatic Randomized Trial. Front Med (Lausanne). 2021 Feb 15;8:605647. doi: 10.3389/fmed.2021.605647. eCollection 2021. PMID 33659261